CLINICAL TRIAL: NCT03381157
Title: Fidgety Movements Analysis in Infants With Cystic Fibrosis
Brief Title: Fidgety Movements in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Akmer Mutlu, Associate Professor, Hacettepe University
Other Study IDs: AkmerMutlu
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cystic Fibrosis
Keywords: general movements, fidgety movements, motor optimality score
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis Group
  Interventions: Other: Observational General Movements Assessments
- Control Group
  Interventions: Other: Observational General Movements Assessments

INTERVENTIONS:
Other: Observational General Movements Assessments — GMs assessment has been increasingly used to predict motor dysfunction, especially the Cerebral Palsy (SP), since its introduction 25 years ago. The GMs assessment is based on the visual holistic perception of normal and abnormal movements of the body. This approach focuses on spontaneous movements of the baby rather than reflexes, tonus, and reactions

SUMMARY:
Very low birth weight infants who are at risk for chronic lung diseases may also be at risk for brain anomalies such as increased echogenicity, leukomalacia and intracranial hemorrhage. Infants with bronchopulmonary dysplasia have been reported to have worse neurodevelopmental outcomes than healthy infants. It has also been pointed out that babies with prolonged and recurrent apneas during sleep may have weak General Movements (GMs) repertoire.

It has been mentioned that motor development retardation may also occur in neurodevelopmental diseases, genetic diseases and chronic lung diseases, as well as in cystic fibrosis. In infants with cystic fibrosis, motor development may be affected by increased incidence of hospitalization, previous infections, malnutrition, respiratory and digestive system disorders. There is no research done with GMs assessment to determine motor dysfunction in infants with cystic fibrosis and this topic is open to research.

Having more information about the motor development of babies by determining the motor characteristics and motor performance of infants with cystic fibrosis, it may be possible to start the disease-specific physiotherapy and rehabilitation programs as early as possible. For this reasons, in the study the investigators aimed to investigate the characteristics of GMs in the "Fidgety" period of 3-5 month term infants diagnosed with cystic fibrosis, to determine the motor performances and to investigate the relation between the GMs characteristics and the features of the disease.

The hypotheses the investigators have set for this study are listed below;

Ho: Spontaneous movements of the "Fidgety" period of infants diagnosed with 3-5 months of cystic fibrosis are not different from normal infants.

H1: Spontaneous movements of "Fidgety" period of infants diagnosed with cystic fibrosis between 3-5 months are different from normal infants.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with cystic fibrosis
* Being between the postterm 3rd and 5th months

Exclusion Criteria:

* Having congenital anomalies,
* Having an ongoing infection,
* Risk of high or low neurological impairment due to perinatal stroke, perinatal asphyxia, intra / peri-ventricular hemorrhage (IVH / PVL), bronchopulmonary dysplasia,
* Fidgety movements evaluation results; being abnormal (AF), sporadic (F +/-) or non-F (F-)
* Baby's family does not want to be involved in the work

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Postterm 3-5 months of cystic fibrosis diagnosed and postterm 3-5 months healthy infants will be included to the study. The number of individuals to be included in the cystic fibrosis group was determined as 19 according to the power analysis at α = 0.05 and β = 0.20 (for 80% power). Within the scope of our study, the control group, which will be formed from postpartum 3-5 month healthy infants, will be composed of our patients who have been taken to the rehabilitation sessions of our clinic on the given days as well as our patients who have been in control for a certain period of time at Hacettepe University Department of Physiotherapy and Rehabilitation, Developmental and Early Physiotherapy Unit, relatives.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Motor Optimality Score (MOS) | 45 minute for each patient
  The MOS has a max. value of 28 (for the best possible performance) and a min. value of 5. The score sheet comprises the following five sub-categories: fidgety movements, age-adequacy of motor repertoire, quality of movement patterns other than fidgety movements, posture, and overall quality of the motor repertoire.
  1. Fidgety Movements; normal fidgety: 12 points, abnormal fidgety: 4 points and sporadic fidgety: 1 points
  2. Age-adequacy of motor repertoire; normal motor repertoire: 4 points, decreased motor repertoire: 2 points, non age-adequacy of motor repertoire: 1 points
  3. Quality of movement patterns other than fidgety movements; normal movement patterns: 4 points, equal normal and abnormal movement patterns: 2 points, abnormal movement patterns: 1 points
  4. Posture; normal posture: 4 points, equal normal and abnormal posture: 2 points, abnormal posture: 1 points
  5. Overall quality of the motor repertoire; normal: 4 points, abnormal: 2 points, cramped-synchronized: 1 points

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Departmant of Pyhsiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herrero D, Einspieler C, Panvequio Aizawa CY, Mutlu A, Yang H, Nogolova A, Pansy J, Nielsen-Saines K, Marschik PB; GenGM Study Group. The motor repertoire in 3- to 5-month old infants with Down syndrome. Res Dev Disabil. 2017 Aug;67:1-8. doi: 10.1016/j.ridd.2017.05.006. Epub 2017 Jun 3. PMID 28586709
- [Background] Einspieler C, Peharz R, Marschik PB. Fidgety movements - tiny in appearance, but huge in impact. J Pediatr (Rio J). 2016 May-Jun;92(3 Suppl 1):S64-70. doi: 10.1016/j.jped.2015.12.003. Epub 2016 Mar 17. PMID 26997356
- See also: Prechtl´s Method on the Qualitative Assessment of General Movements — http://general-movements-trust.info